CLINICAL TRIAL: NCT00000964
Title: The Effect of Increasing Gastric pH Upon the Bioavailability of Orally Administered Phosphonoformic Acid (Foscarnet)
Brief Title: The Effect of Stomach Acid on Foscarnet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 136; 11111 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Ranitidine; Phosphorus Acids; Drug Evaluation; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ranitidine; Foscarnet

INTERVENTIONS:
Drug: Ranitidine hydrochloride
Drug: Foscarnet sodium

SUMMARY:
To see if ranitidine, by reducing stomach acidity, can enhance the effectiveness of foscarnet, by making foscarnet more available to the body.

Foscarnet is an antiviral compound. Laboratory studies have shown it to be active against HIV. However, only 12 - 22 percent of an oral foscarnet dose is absorbed by the body. Ranitidine suppresses gastric acid output, increasing gastric pH. Thus by increasing gastric pH (decreasing stomach acidity), less foscarnet is expected to be decomposed or broken down in the stomach. Thus, more foscarnet should be absorbed into the body.

DETAILED DESCRIPTION:
Foscarnet is an antiviral compound. Laboratory studies have shown it to be active against HIV. However, only 12 - 22 percent of an oral foscarnet dose is absorbed by the body. Ranitidine suppresses gastric acid output, increasing gastric pH. Thus by increasing gastric pH (decreasing stomach acidity), less foscarnet is expected to be decomposed or broken down in the stomach. Thus, more foscarnet should be absorbed into the body.

Six asymptomatic HIV-infected males, or those with limited symptoms of early AIDS-related complex ( ARC ), will receive one dose intravenously of ranitidine in distilled water and one dose of placebo (distilled water alone), followed in 1 hour by foscarnet in oral solution. The order of ranitidine and placebo is randomized and the two foscarnet doses are separated by at least 72 hours. A nasogastric pH probe is placed on each morning of drug administration to monitor gastric pH.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acetaminophen and sedatives.

Patient must be able to give informed consent.

Exclusion Criteria

Patients with the following are excluded:

* Unintentional weight loss in excess of 10 pounds or 10 percent of usual body weight within 2 years prior to study.
* Unexplained temperature above 38 degrees Celsius on more than 5 consecutive days or on more than 10 days in any 30 days in 2 years prior to expected study entry.
* Unexplained diarrhea defined by two or more stools/day for at least 14 days during a 120-day interval.

Prior Medication:

Excluded within 1 week of entry into study:

* Probenecid, aspirin, or diuretics.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Study Completion 1990-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DM Kornhauser, Study Chair
Locations (1):
- Johns Hopkins Adult AIDS CRS, Baltimore, Maryland, United States

REFERENCES:
- [Background] Barditch-Crovo PA, Petty BG, Gambertoglio J, Nerhood LJ, Kuwahara S, Hafner R, Lietman PS, Kornhauser DM. The effect of increasing gastric pH upon the bioavailability of orally-administered foscarnet. Antiviral Res. 1998 Jun;38(3):209-12. doi: 10.1016/s0166-3542(98)00024-2. PMID 9754889